CLINICAL TRIAL: NCT01015573
Title: Database Creation and Evaluation of Motor Function of Finger Tapping Measured by Magnetic Sensor System in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Fumiko Higashikawa, Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: eki-188
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy subjects (Experimental)
  Interventions: Device: magnetic sensor system to measure the movements of finger tapping

INTERVENTIONS:
Device: magnetic sensor system to measure the movements of finger tapping

SUMMARY:
The purpose of this study is to create a database of quantified finger movements. Using the evaluation system with magnetic sensors, the movements of finger tapping are measured and assessed by various indices, such as finger tapping interval, maximum amplitude of finger taps, and so on. In this study, the investigators will accumulate the data from healthy subjects for the purpose of applying this evaluation system to diagnosis support of nervous diseases in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Informed consent signed

Exclusion Criteria:

* Renal or hepatic dysfunction
* Severe heart disease
* Under medications for diabetes or hypertension
* Medical history of nervous disease, mental disease, muscular disease, cervical spondylosis, and/or apoplexy
* Feeling difficulty in daily movements
* Taking medicines which possibly affect the motor function of finger tapping.
* Implantation of pacemaker or DBS

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
movements of finger tapping | 1 day for measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan